CLINICAL TRIAL: NCT04143334
Title: Prevalence of Blindness, Visual Impairment and Main Avoidable Causes in Chao Nan Area
Brief Title: Prevalence of Blindness, Visual Impairment in Chao Nan Area, China
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, ZHANG XIUJUAN, Dr. Principal Investigator, Chinese University of Hong Kong
Other Study IDs: CRE-2011.389
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Blindness; Cataract; Visual Impairment; Refractive Errors
Keywords: blindness; cataract blindness; diagnostic accuracy
MeSH Terms: conditions — Blindness; Cataract; Vision Disorders; Refractive Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RAAB survey: We will examine 3700 Chaonan County residents aged 50 years and older, selected via a clustered, randomized sampling with probability proportional to size (PPS). The cluster will be at the village level, 50 subjects aged 50 years and older will be examined in each cluster includes Visual acuity, torch light, and fundus review, the major cause of blindness or visual impairment will be determined.
  Interventions: Diagnostic Test: Conventional survey
- conventional survey: All the recruited participants underwent ophthalmic examination according to the RAAB protocol and then 60% of them were re-examined with instruments in a mobile eye clinic set up in a village center on the same day. Examination in the mobile clinic included standardized visual acuity (VA) tests using logarithm of the minimum angle resolution charts, refraction, slit-lamp biomicroscopy, and dilated fundal examination with a binocular indirect ophthalmoscope.
  Interventions: Diagnostic Test: Conventional survey

INTERVENTIONS:
Diagnostic Test: Conventional survey

SUMMARY:
This study will provide a profile of blindness/visual impairment, avoidable blindness and cataract surgery service in Chaonan, mainland China. We also evaluate the diagnostic accuracy of Rapid Assessment of Avoidable Blindness (RAAB) comparison with conventional survey.

DETAILED DESCRIPTION:
This proposal describes a population-based study aimed at determining the prevalence of visual impairment, blindness and major causes in adults age 50 years old and above in Chaonan County of Guangdong province, where one of the Project Vision Charity Eye center was founded in 2009.

In the proposed study, we will examine 3700 Chaonan County residents aged 50 years and older, selected via a clustered, randomized sampling with probability proportional to size (PPS). The cluster will be at the village level, 50 subjects aged 50 years and older will be examined in each cluster includes Visual acuity, torch light, and fundus review, the major cause of blindness or visual impairment will be determined. We also randomly recruited 60% clusters,total 2250 participants, from RAAB survey to conduct a detailed conventional eye examination.

This study will provide a profile of blindness/visual impairment, avoidable blindness and cataract surgery service in Chaonan. we will evaluate the diagnostic accuracy of Rapid Assessment of Avoidable Blindness (RAAB) comparison with conventional survey. . It will provide important public health issues for the purposes of establishing a sustainable and suitable model to eliminate the cataract blindness in China.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 years and above
* In each household all persons , residing in the household for six months or more over the past year
* "Residing in the household" is defined as "sharing meals from the same kitchen with the other members of the household for at least 6 months in a year. Exclude any visitors.

Exclusion Criteria:

* age <50 years old
* Visitors in the villages
* Residing in the household< 6 months

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Among the 3700 people, 169 (4.6%) could not be reached, 20 (0.5%) were unable to communicate, and 27 (0.7%) refused. Consequently, 3484 persons (response rate 94.2%) with a mean (±SD) age of 64.4±9.8 years were examined. These included 1397 men (40.1%) with an average age of 65.3 ±9.6 years and 2087 women (59.9%) with an average age of 63.8±9.8 years.
  Of the 2145 subjects (95.3%，2145/2250), 327 (15.2%) refused, and 2 (0.1%) were unable to cooperate for examination. Consequently, 1816 subjects (1816/2145, 84.7%) with a mean (±SD) age of 64.4±9.6 years received the conventional ophthalmic examination in the mobile eye clinic (figure 1). These included 686 men (37.8%) with an average age of 65.5±9.4 years and 1130 women (62.2%) with an average age of 63.8±9.6 years.
Sampling Method: Probability Sample
Enrollment: 3700 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
the prevalence of blindness and visual impairment (VI) and main avoidable causes in Chaonan, China | one year
  the prevalence of blindness and visual impairment (VI), and report the avoidable causes, including cataract in Chaonan Region, Guangdong Province, southern China

SECONDARY OUTCOMES:
the diagnostic accuracy of RAAB | one year
  To evaluate the diagnostic accuracy of Rapid Assessment of Avoidable Blindness (RAAB)

CONTACTS AND LOCATIONS:
Overall Officials: XIUJUAN ZHANG, PhD, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li EY, Liu Y, Zhan X, Liang YB, Zhang X, Zheng C, Jhanji V, Xu P, Chang DF, Lam DS. Prevalence of blindness and outcomes of cataract surgery in Hainan Province in South China. Ophthalmology. 2013 Nov;120(11):2176-83. doi: 10.1016/j.ophtha.2013.04.003. Epub 2013 May 25. PMID 23714323